CLINICAL TRIAL: NCT06467838
Title: Airway Approaches of Anesthesiology and Reanimation Physicians in Cervical Neck Trauma Patients in Turkey: A Survey Study
Brief Title: Airway Approaches of Anesthesiology and Reanimation Physicians in Cervical Neck Trauma Patients in Turkey
Status: Active, not recruiting | Type: Observational
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Collaborators: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, EMİNE YURT, Medical Doctor, Kocaeli Derince Education and Research Hospital
Other Study IDs: 2023-48
Record Dates: First submitted 2024-06-03; First posted 2024-06-21 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Trauma Patients; Surgery; Trauma; Survey
Keywords: DIFFICULT AIRWAY; CERVICAL NECK TRAUMA; A SURVEY STUDY
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Title: Airway Approaches of Anesthesiology and Reanimation Physicians in Cervical Neck Trauma Patients in Turkey: A Survey Study This study aims to evaluate the knowledge, awareness levels, and equipment adequacy of anesthesiology and reanimation physicians in Turkey regarding airway management in cervical neck trauma patients through a 32-question online survey. The findings will inform targeted improvements in training and resource allocation to enhance clinical outcomes in this patient population.

DETAILED DESCRIPTION:
Airway Approaches of Anesthesiology and Reanimation Physicians in Cervical Neck Trauma Patients in Turkiye

The management of airway in patients with cervical neck trauma presents unique challenges due to the associated difficulty in ventilation, intubation, and potential complications. Airway-related issues are a critical determinant of morbidity and mortality in this patient population. This study aims to evaluate the current practices and perspectives of anesthesiology and reanimation physicians in Turkey regarding airway management in cervical neck trauma cases.

The primary objective of this survey-based study is to assess the techniques and methods employed by anesthesiology and reanimation physicians in the airway management of cervical neck trauma patients.

The study aims to:

Investigate the variability in airway management approaches. Identify the equipment used during intubation. Determine the need for additional training in airway management for these patients.

Examine how well the practical applications align with the algorithms specified in the "Difficult Airway Management Guidelines".

This study will be conducted using a structured survey developed on the Google Forms platform, comprising three sections:

Consent: Participants will be asked if they consent to participate in the survey.

Demographic Data: Collection of basic demographic information about the participants.

Airway Management Practices: A comprehensive set of 32 questions using multiple-choice, checkboxes, and open-ended formats to gather detailed information on the airway management approaches and intubation techniques used in patients with cervical trauma.

The insights gained from this survey will provide valuable data on the current practices of anesthesiology and reanimation physicians in Turkey, highlighting areas where additional training may be required. Understanding these practices can help guide the development of improved protocols and training programs to ensure safer airway management and anesthesia practices in patients with cervical neck trauma. This study aims to contribute to the optimization of clinical outcomes by aligning practical approaches with established guidelines for difficult airway management.

By evaluating the current state of airway management in cervical neck trauma patients, this study will offer guidance on necessary precautions and training to enhance patient safety and reduce complications. The findings will help inform clinical practice and policy, fostering a multidisciplinary approach to the management of these high-risk patients.

Cervical spine trauma encompasses a variety of injuries, from minor muscle strains to life-threatening fracture-dislocations associated with spinal cord lesions. Endotracheal intubation carries significant risks in patients with cervical fractures. Hyperextension of the neck can cause spinal cord injury. In the evaluation and management of cervical trauma patients, airway safety and cervical spine stabilization should be ensured first. Inappropriate airway management in patients with cervical spine injuries can have adverse effects on neurological damage. In cervical trauma patients, especially during intubation, head and neck movement can be minimized by stabilizing the head with a neck collar, if necessary. Mobility of the cervical spine may lead to decreased laryngeal vision and unsuccessful intubation during laryngoscopy.

Various tools and methods can be used to provide airway access in cervical trauma patients. Intubation with various airway devices causes extension of the cervical spine. It is anticipated that mask ventilation may be difficult for patients who receive anesthesia and/or muscle relaxants for intubation, and if the first attempts at intubation are unsuccessful, a hypoxic condition will be encountered. The main concern of anesthesiologists in airway management in cervical trauma patients is to avoid prolonged intubation and excessive cervical movement. No technique for airway management has been reported to be superior to others for preventing neurological deterioration in patients with unstable cervical spine. The technique chosen depends on the clinic situation, patient factors, and the experience of the clinician. In short, in patients with an unstable cervical spine, anesthesiologists should keep in mind that there may be neurological deficits during laryngoscopy, the possibility of difficult intubation, and that the neck should be moved as little as possible, with or without a cervical collar.

Various intubation techniques are used in cervical trauma patients, depending on the availability of airway equipment and the experience of the anesthesiologist. These include techniques such as direct laryngoscopy and intubation, video laryngoscopy and intubation, awake fiberoptic intubation, and aintree catheter-mediated fiberoptic intubation via LMA. Fiberoptic intubation, which minimizes cervical spine movement, is considered the more preferred method in these patients, and its success rate varies between 50% and 90%. However, the success rate of intubation may decrease in some cases, such as the presence of a patient who cannot cooperate with the anesthetist and the presence of blood and secretions in the patient's airway.

Extubation of patients with cervical trauma is important. The decision to extubate is an important decision to be made according to the scope of the surgery, the time of the operation, the patient's accompanying pathologies and the complications of the operation. If any questions about the airline come to mind; The patient should not be extubated until the patient is fully awake, obeys verbal commands, and is determined to maintain the airway safely. Edema, bleeding that may occur in the neck and airway, and plates placed on the neck may make a new intubation more difficult. We planned to evaluate this issue through the questions in our survey.

You can access our work from the link below:

Links: http://docs.google.com/forms/d/1aQSbby6Vi2-qdJIakiklWeQYCrIY3Kk8jZicxEMqOKw/edit

ELIGIBILITY:
Inclusion Criteria:

* Becoming an Anesthesiology and Reanimation physician

Exclusion Criteria:

* Those who are not an anesthesiologist or reanimation physician are excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The data collection tool in the research is a survey. The scope of the research consists of anesthesia and reanimation physicians. The survey form consists of three parts. In the first part, they will be asked whether they will participate in the survey. In the second section, descriptive questions regarding the demographic characteristics of the participants were included. In the third section, questions to measure airway approaches to cervical neck trauma patients are included.
Sampling Method: Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Survey | 6 months
  Knowledge and Awareness Level:Assessment of the baseline knowledge and awareness levels of anesthesiology and reanimation physicians in Turkey regarding the airway management of cervical neck trauma patients.
SURVEY | 6 months
  Evaluation of the availability and adequacy of the equipment used by physicians during airway management in cervical neck trauma cases. This measure will determine whether the existing equipment meets the standards required for safe and effective intubation and ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: EMINE YURT, Principal Investigator — Kocaeli Derince Education and Research Hospital
Locations (1):
- KocaeliDERH, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Airway Approaches of Anesthesiology and Reanimation Physicians in Cervical Neck Trauma Patients in Turkey: A Survey Study — http://docs.google.com/forms/d/1aQSbby6Vi2-qdJIakiklWeQYCrIY3Kk8jZicxEMqOKw/edit